CLINICAL TRIAL: NCT06402617
Title: Ablation of Focal Activation During Persistent Atrial Fibrillation to Determine the Characteristics of Focal Drivers
Brief Title: Ablation of Focal Activation in Atrial Fibrillation
Acronym: RETRO-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22HH8087; IRAS Project ID: 328297 (Other: UK Integrated Research Application System)
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Persistent; Arrhythmia; Arrhythmias, Cardiac; Cardiac Arrhythmia
Keywords: ablation; electrophysiology; mapping; local activation time; pulmonary vein isolation; atrial fibrillation cycle length
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: This will be a single-centre pilot study that will take place over 36 months. We will randomise 110 participants, half to a control arm that receives standard clinical care, and half to a treatment arm that receives the same care alongside adjunctive ablation of sites of focal activation identified by RETRO-Mapping. Both arms will also undergo additional intraprocedural measurements using RETRO-Mapping, and atrial fibrillation cycle length with standard tools. Randomisation will be by block randomisation for each site by closed envelope in sets of 10 containing five control arm and five test arm allocations.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to their treatment group, and outcomes will be studied prospectively on both an intention-to-treat and a per-protocol basis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation with diagnostic RETRO-Mapping only (Placebo Comparator): All patients will undergo standard pulmonary vein isolation (PVI) procedures with 3D electroanatomic mapping using the CARTO™ system (Biosense Webster, USA), or the EnSite X™ system (Abbott, USA). A decapolar catheter will be inserted into the coronary sinus. A 3D electroanatomic map of the left atrium will be created and all pulmonary veins will be identified. Radio-frequency ablation will be performed to achieve PVI.
  After the PVI procedure, patients in the control arm will have the same mapping for identification and categorisation of focal sources, but no adjunctive ablation. RETRO-Mapping will be performed using custom-built hardware called Tau20 that has been validated for reproducibility against existing commercial technologies.
  Interventions: Procedure: Pulmonary vein isolation; Diagnostic Test: RETRO-Mapping without adjunctive ablation
- Pulmonary vein isolation with adjunctive ablation guided by RETRO-Mapping (Experimental): In addition to and after the PVI procedure, patients the intervention arm will then have RETRO-Mapping performed of the remaining atria and atrial fibrillation cycle length measured in coronary sinus and left atrial appendage. Each segment will be mapped for 30 seconds and the activation pattern categories; if focal activation is identified, it will then be ablated. A further 30 seconds will be mapped at the same segments post-ablation to determine effect. The coronary sinus and left atrial appendage cycle length will be documented at the start of RETRO-Mapping and after each lesion set.
  Interventions: Procedure: Pulmonary vein isolation; Procedure: Adjunctive ablation guided by RETRO-Mapping

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Standard clinical radio-frequency ablation isolation of pulmonary veins
Diagnostic Test: RETRO-Mapping without adjunctive ablation — RETRO-Mapping performed using research equipment and software, but without any adjunctive ablation
  Arms: Pulmonary vein isolation with diagnostic RETRO-Mapping only
Procedure: Adjunctive ablation guided by RETRO-Mapping — Radio-frequency ablation using a European conformity (CE)-marked ablation catheter of sites of focal activation identified by RETRO-Mapping
  Arms: Pulmonary vein isolation with adjunctive ablation guided by RETRO-Mapping

SUMMARY:
Recurrent focal electrical activation (or ectopy) superseding sinus activation is the only mechanism proven to drive paroxysmal atrial fibrillation (AF). However, it has not been possible to show similar focal drivers during AF, owing to the limitations of mapping in persistent AF. RETRO-Mapping has been developed as a method to generate activation maps during AF to test the hypothesis that persistent AF is also maintained by focal drivers.

RETRO-Mapping is able to locate sites of focal activation that were isolated, intermittent, or recurrent during persistent AF. However, a 30-second segment of AF can have approximately 150 wavefronts in a small area of myocardium. Screening for focal activation and manually validating these prior to ablation was not feasible using current commercial systems.

RETRO-Mapping can automatically detect focal activation and a recording system that enables the intracardiac signals to be directly analysed by the RETRO-Mapping software. This will allow RETRO-Mapping to build a detailed classification of focal activation types and study the impact of ablation of these sites on the AF cycle length, to address the hypothesis that persistent AF is maintained by focal drivers.

DETAILED DESCRIPTION:
Multiple large, prospective randomised controlled trials have shown that pulmonary vein isolation (PVI) terminates AF in 50-70% of cases. The continued presence of atrial fibrillation (AF) in those without demonstrable reconnection on a mapping catheter suggests other mechanisms at play. However, outside PV ectopy, drivers of AF initiation or maintenance remain unclear.

Detailed mapping studies have confirmed the presence of both focal activation and spatiotemporally stable planar wavefronts during AF, with limited data suggesting focal activation may drive AF. This study is based on the hypothesis that focal activation may lead to planar wavefronts at its origin, which subsequently disintegrate on exposure to refractory myocardium in different locations, and assumes that randomised studies of adjunctive ablation have shown poor results to date because excessive ablation has been performed at non-driver sites and this ablation scar is pro-arrhythmic.

RETRO-Mapping is a novel algorithmic solution to AF mapping with published validation confirming accuracy of analysis of activation wavefronts, when benchmarked against laborious manual annotation. RETRO-Mapping found that nearly 30% of mapped sites contained focal activation, and these ranged from single events to repetitive events that could either be consecutive or interspersed with other activation patterns. This study now aims to characterise multiple different activation patterns that exist within the milieu of AF, and interrogate their role in the initiation and maintenance of AF by randomising patients to adjunctive ablation of sites of focal activation, versus usual care alone (i.e., PVI).

The effect of this adjunctive ablation on AF cycle length will be the primary outcome measure, and freedom from AF will be a secondary outcome measure. AF termination is usually considered a positive endpoint for adjunctive ablation, but, as a single event, cannot help identify which part of the adjunctive ablation approach led to this useful outcome. By contrast, left atrial appendage and coronary sinus cycle length prolongation can be used as continuous measures of progress towards AF termination, and may allow determination of whether focal activation sites are drivers of persistent AF, and whether the characteristics of focal activation alter the likelihood of it being a driver.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation with clinical indication for catheter ablation
* Clinically suitable candidate for catheter ablation
* Signed informed consent

Exclusion Criteria:

* Previous atrial fibrillation or other catheter ablation procedure
* Clinical contraindication to catheter ablation or general anaesthetic, including history of adverse reaction to contrast media, or presence of intracardiac thrombus, or inadequate anticoagulation in the preceding 6 weeks
* Valvular disease graded moderate or greater, or presence of a prosthetic valve
* Moderate-to-severe heart failure, defined as left ventricular ejection fraction <35% and/or New York Heart Association class III-IV
* Any form of cardiomyopathy
* Active infection or fever
* Severe cerebrovascular disease
* Active gastrointestinal bleeding
* Bleeding or clotting disorders, clinically high bleeding risk, or clinical contraindication to receiving heparin
* Baseline serum creatinine >200umol/L
* Currently receiving or at risk of requiring renal replacement therapy
* Uncontrolled diabetes (HbA1c ≥73mmol/mol or HbA1c ≤64mmol/mol and fasting blood glucose ≥9.2mmol/L)
* Malignancy necessitating therapy
* Life expectancy shorter than the duration of the trial
* Pregnancy, or childbearing potential and not using a highly effective method of contraception
* Inability to provide informed consent to participate in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation cycle length in coronary sinus and left atrial appendage | Intra-procedural
  Measurement of atrial fibrillation cycle length in coronary sinus and left atrial appendage, measured in miliseconds

SECONDARY OUTCOMES:
Freedom from atrial fibrillation | 1 year
  Follow-up after a 3-month blanking period. Recurrence of atrial arrhythmia at 3, 6, 9, and 12 months with a 24-hour Holter monitor, or at any point over same period with an AliveCor KardiaMobile, will be recorded. Measurements across differing devices will be aggregated to give a single time-to-recurrence measurement, given in days.

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, FRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No